CLINICAL TRIAL: NCT00606736
Title: Relativity Study Between Idiopathic Ventricular Arrhythmia and Sex Hormone Levels in Different Stages of Menstrual Cycle
Status: Withdrawn | Type: Observational
Why Stopped: it's difficult to recruit enough participants eligible for this study
Sponsor: Harbin Medical University (Other)
Responsible Party: Bai Xiaopeng, Vasculocardiology Deparment ,The Fourth Hospital of Harbin Medical University
Other Study IDs: HMU-007; HMU-008
Record Dates: First submitted 2008-01-22; First posted 2008-02-04 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2008-01

CONDITIONS: Ventricular Premature Complexes
Keywords: right ventricular outflow tract arrhythmia; sex hormone level; menstrual cycle; Gonadal Hormones
MeSH Terms: conditions — Ventricular Premature Complexes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- patients: subjects with right ventricular outflow tract arrhythmia
- control: subjects ,age match,healthy

SUMMARY:
The purpose of this study is to determine whether the occurrence of idiopathic right ventricular outflow tract(RVOT) arrhythmia is relative to sex hormone levels in different stages of female menstrual cycle

DETAILED DESCRIPTION:
The predilection site of idiopathic ventricular arrhythmia is right ventricular outflow tract ,which is called idiopathic RVOT arrhythmia , a retrospective study reported the females are susceptibility to this kind of arrhythmia and another questionaire survey of triggers for RVOT-VT initiation indicated that women have RVOT-A initiation with recognized states of sex hormonal flux , but few researches were made to study the exact relation between this kind of arrhythmia and sex hormone levels, this is the aim of our study .40 females with regular menses(20 females with RVOT arrhythmia ,20 healthy volunteers) will be screened, the Participants will undergo ECG monitoring and their blood samples will be collected at various times throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Must be female
* Aged 20 to 45 years, with regular menstrual cycles.
* With normal BMI
* Without organic heart disease
* Healthy volunteers and women with RVOT arrhythmia are both being recruited.

Exclusion Criteria:

* Pregnancy
* Use of hormonal therapy including birth control pills or other drugs

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women aged 20 to 45 years with regular menstrual cycles.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
number and duration of right ventricular outflow tract arrhythmia | one month

SECONDARY OUTCOMES:
sex hormone levels | one month

CONTACTS AND LOCATIONS:
Overall Officials: Xueqi Li, doctor, Study Director — the fourth hospital of harbin medical university
Locations (1):
- Cardiology Department of the 4Th Hospital of Harbin Medical University, Harbin, Heilongjiang, China